CLINICAL TRIAL: NCT00847145
Title: A Phase 3, Open Label, Multi-Center, Extension Study to Evaluate the Safety, Tolerability and Immunogenicity of Novartis Meningococcal B Recombinant Vaccine When Administered as a Booster at 12 Months of Age or as a Two-dose Catch-up to Healthy Toddlers Who Participated in Study V72P13
Brief Title: Extension Study of V72P13 to Evaluate the Safety, Tolerability and Immunogenicity of Novartis Meningococcal B Recombinant Vaccine When Administered as a Booster or as a Two-dose Catch-up to Healthy Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V72P13E1; 2008-006301-17 (EudraCT Number)
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Meningococcal Disease
Keywords: toddler; Meningococcal disease; prevention; vaccination
MeSH Terms: conditions — Meningococcal Infections

ARMS (8):
- 12B12M (1a) (Experimental): Previously in the parent study subjects had received three doses of rMenB+OMV NZ and routine vaccine at 2, 4 and 6 months of age,respectively. These subjects received a booster (fourth) dose at 12 months of age concomitantly with one dose of MMRV vaccine in the present study.
  Interventions: Biological: 1a - rMenB+OMV NZ and routine vaccines
- 12B13M (1b) (Experimental): Previously in the parent study subjects had received three doses of rMenB+OMV NZ and routine vaccine at 2, 4 and 6 months of age, respectively. These subjects received a booster (fourth) dose at 12 months and one dose of MMRV vaccine at 13 months of age in the present study.
  Interventions: Biological: 1b - rMenB+OMV NZ and routine vaccines
- 12M13B15B (2a) (Experimental): Previously in the present study subjects had received routine vaccine at 2, 4 and 6 months of age respectively. These subjects received MMRV vaccine at 12 months of age and two catch-up doses of rMenB+OMV NZ vaccine at 13 and 15 months of age in the present study.
  Interventions: Biological: 2a - Routine and rMenB+OMV NZ vaccines
- 12M12B14B (2b) (Experimental): Previously in the parent study subjects ahd received three doses of routine vaccine at 2, 4 and 6 months of age, respectively. These subjects received two catch-up doses of rMenB+OMV NZ at 12 and 14 months of age and one dose of MMRV vaccine given concomitantly at 12 months of age in the present study.
  Interventions: Biological: 2b - rMenB+OMV NZ and routine vaccines
- 12B12M (3a) (Experimental): Previously in the parent study subjects had received three doses of rMenB+OMV NZ at 2, 4 and 6 months of age respectively. These subjects had received one booster (fourth) dose of rMenB+OMV NZ at 12 months of age concomitantly with one dose of MMRV vaccine in the present study.
  Interventions: Biological: 3a - rMenB+OMV NZ and routine vaccines
- 12B13M (3b) (Experimental): Previously in the present study subjects had received three doses of rMenB+OMV NZ at 12 months of age respectively. These subjects one booster (fourth) dose of rMenB+OMV NZ at 12 months of age and one dose of MMRV vaccine at 13 months of age in the present study.
  Interventions: Biological: 3b - 1 dose of rMenB+OMV NZ plus routine infant vaccinations
- 12B12M_C (4a) (Experimental): Previously in the parent study subjects had received three doses of Meningococcal C vaccine and routine vaccine at 2, 4 and 6 months of age respectively. These subjects had received one single dose of rMenB+OMV NZ at 12 months of age concomitantly with one dose of MMRV vaccine in the present study.
  Interventions: Biological: 4a- rMenB+OMV NZ and routine vaccines
- 12B13M_C (4b) (Experimental): Previously in the parent study subjects had received three doses of Meningococcal C vaccine and routine vaccine at 2, 4 and 6 months of age. These subjects received one single dose o rMenB+OMV NZ at 12 months of age and one dose of MMRV vaccine at 13 months of age in the present study.
  Interventions: Biological: 4b - rMenB+OMV NZ and routine vaccines

INTERVENTIONS:
Biological: 1a - rMenB+OMV NZ and routine vaccines — One dose of rMenB vaccine and routine vaccine at study month 12.
  Arms: 12B12M (1a)
Biological: 1b - rMenB+OMV NZ and routine vaccines — One dose of rMenB vaccine at study month 12 and routine vaccine at study month 13.
  Arms: 12B13M (1b)
Biological: 2a - Routine and rMenB+OMV NZ vaccines — One dose of routine vaccine at study month 12 and two doses of rMenB vaccine at study months 13 and 15.
  Arms: 12M13B15B (2a)
Biological: 2b - rMenB+OMV NZ and routine vaccines — Two doses of rMenB vaccine at study months 12 and 14 and one dose of routine vaccine at study month 12.
  Arms: 12M12B14B (2b)
Biological: 3a - rMenB+OMV NZ and routine vaccines — One dose of rMenB vaccine and one dose of routine vaccine at study month 12.
  Arms: 12B12M (3a)
Biological: 3b - 1 dose of rMenB+OMV NZ plus routine infant vaccinations — One dose of rMenB vaccine at study month 12 and one dose of routine vaccine study month 13.
  Arms: 12B13M (3b)
Biological: 4a- rMenB+OMV NZ and routine vaccines — One dose of rMenB vaccine and one dose of routine vaccine at study month 12.
  Arms: 12B12M_C (4a)
Biological: 4b - rMenB+OMV NZ and routine vaccines — One dose of rMenB vaccine and one dose of routine vaccine at study month 12.
  Arms: 12B13M_C (4b)

SUMMARY:
The proposed study is an Extension Study of V72P13 to Evaluate the Safety, Tolerability and Immunogenicity of Novartis Meningococcal B Recombinant Vaccine When Administered as a Booster at 12 Months of Age or as a Two-dose Catch-up to Healthy Toddlers

ELIGIBILITY:
Inclusion Criteria:

* Healthy 12-month-old toddlers (0/ +29 days) who completed Study V72P13

Exclusion Criteria:

* Previous ascertained or suspected disease caused by N. meningitidis;
* History of severe allergic reaction after previous vaccinations or hypersensitivity to any vaccine component;
* Any serious chronic or progressive disease
* Known or suspected impairment/ alteration of the immune system,
* Receipt of, or intent to immunize with another vaccine, within 30 days prior to enrollment.

Ages: 365 Days to 394 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2249 (Actual)
Dates: Start 2009-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (59):
- Austria (7):
  - Altenburger, Eisenstadt
  - Grässl, Hall in Tirol
  - Häckel, Kirchdorf
  - Prieler, Neufeld A.d. Leitha
  - Maurer, Salzburg
  - Sommer, Vienna
  - Angermayr, Wels
- Czechia (16):
  - Site 27, Boskovice
  - Site 19, Brno
  - Site 22, Chomutov
  - Site 12, Havlíčkův Brod
  - Fakulta vojenskeho zdravotnictví, Hradec Králové
  - Site 28, Hranice I-mesto
  - Site 13, Humpolec
  - Site 25, Kladno
  - Site 21, Kolín
  - Site 10, Liberec
  - Site 24, Litoměřice
  - Site 17, Ostrava
  - Site 18, Ostrava-Poruba
  - Site 16, Pilsen
  - Site 26, Rumburk
  - Site 23, Ústí nad Labem
- Finland (15):
  - Site 30, Espoo
  - Site 31, Helsinki
  - Site 32, Helsinki
  - Site 34, Jarvenpaa
  - Site 35, Kokkola
  - Site 45, Kotka
  - Site 46, Kuopio
  - Site 47, Lahti
  - Site 49, Oulu
  - Site 50, Pori
  - Site 51, Seinäjoki
  - Site 52, Tampere
  - Site 53, Turku
  - Site 33, Vantaa
  - Site 48, Vantaa
- Germany (14):
  - Site 99, Detmold
  - Site 92, Espelkamp
  - Site 95, Freising
  - Site 64, Fulda
  - Site 58, Lauffen am Neckar
  - Site 57, Marbach A. N.
  - Site 80, München
  - Site 83, München
  - Site 97, München
  - Site 96, München
  - Site 91, Műnchen
  - Site 81, Porta Westfalica
  - Site 65, Schwieberdingen
  - Site 94, Weilheim
- Italy (7):
  - Dipartimento di Scienze della Salute, Genova, Genova
  - Fondazione IRCCS Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena Italia, Milan, Milano
  - Pediatria dell' Ospedale Sacco, Milan, Milano
  - Istituto di Igiene e Medicina Preventiva - Università degli Studi di Sassari, Sassari, Sassari
  - ASL/TA, Taranto, Taranto
  - Universita degli Studi di Messina, Policlinico G. Martino, Messina
  - Ospedale Maggiore di Novara, Novara

REFERENCES:
- [Derived] Zafack JG, Bureau A, Skowronski DM, De Serres G. Adverse events following immunisation with four-component meningococcal serogroup B vaccine (4CMenB): interaction with co-administration of routine infant vaccines and risk of recurrence in European randomised controlled trials. BMJ Open. 2019 May 19;9(5):e026953. doi: 10.1136/bmjopen-2018-026953. PMID 31110098
- [Derived] Vesikari T, Esposito S, Prymula R, Ypma E, Kohl I, Toneatto D, Dull P, Kimura A; EU Meningococcal B Infant Vaccine Study group. Immunogenicity and safety of an investigational multicomponent, recombinant, meningococcal serogroup B vaccine (4CMenB) administered concomitantly with routine infant and child vaccinations: results of two randomised trials. Lancet. 2013 Mar 9;381(9869):825-35. doi: 10.1016/S0140-6736(12)61961-8. PMID 23324563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 15 sites in Finland, 12 sites in Germany, 5 sites in Austria, 27 sites in Czech Republic and 6 sites in Italy.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- 12B12M (1a): Previously in the parent study (NCT00657709) subjects had received three doses of rMenB+OMV NZ and routine vaccine at 2, 4 and 6 months of age, respectively. These subjects received a booster (fourth) dose at 12 months of age concomitantly with one dose of MMRV vaccine in the present study.
- 12B13M (1b): Previously in the parent study (NCT00657709) subjects had received three doses of rMenB+OMV NZ and routine vaccine at 2, 4 and 6 months of age, respectively. These subjects received a booster (fourth) dose at 12 months and one dose of MMRV vaccine at 13 months of age in the present study.
- 12M12B14B (2b): Previously in the parent study (NCT00657709) subjects had received three doses of routine vaccine at 2, 4 and 6 months of age, respectively. These subjects received two catch-up doses of rMenB+OMV NZ at 12 and 14 months of age and one dose of MMRV vaccine given concomitantly at 12 months of age in the present study.
- 12B12M (3a): Previously in the parent study (NCT00657709) subjects had received three doses of rMenB+OMV NZ at 2, 4 and 6 months of age respectively. These subjects had received one booster (fourth) dose of rMenB+OMV NZ at 12 months of age concomitantly with one dose of MMRV vaccine in the present study.
- 12B12M_C (4a): Previously in the parent study (NCT00657709) subjects had received three doses of Meningococcal C vaccine and routine vaccine at 2, 4 and 6 months of age respectively. These subjects had received one single dose of rMenB+OMV NZ at 12 months of age concomitantly with one dose of MMRV vaccine in the present study.
- 12B13M_C (4b): Previously in the parent study (NCT00657709) subjects had received three doses of Meningococcal C vaccine and routine vaccine at 2, 4 and 6 months of age. These subjects received one single dose of rMenB+OMV NZ at 12 months of age and one dose of MMRV vaccine at 13 months of age in the present study.
Period: Overall Study
Arm/Group | 12B12M (1a) | 12B13M (1b) | 12M13B15B (2a) | 12M12B14B (2b) | 12B12M (3a) | 12B13M (3b) | 12B12M_C (4a) | 12B13M_C (4b)
Started | 629 | 633 | 285 | 117 | 137 | 156 | 152 | 140
Completed | 623 | 627 | 274 | 116 | 131 | 152 | 143 | 136
Not Completed | 6 | 6 | 11 | 1 | 6 | 4 | 9 | 4
Not completed — AE or Death | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 6 | 1 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 3 | 1 | 1 | 0 | 4 | 4 | 8 | 2
Not completed — Inappropriate enrollment | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 12B12M (1a) | 12B13M (1b) | 12M13B15B (2a) | 12M12B14B (2b) | 12B12M (3a) | 12B13M (3b) | 12B12M_C (4a) | 12B13M_C (4b) | Total
Number analyzed (Participants) | 629 | 633 | 285 | 117 | 137 | 156 | 152 | 140 | 2249
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.3 (0.5) | 12.3 (0.5) | 12.3 (0.5) | 12.3 (0.5) | 12.2 (0.5) | 12.2 (0.4) | 12.2 (0.5) | 12.2 (0.4) | 12.3 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 290 | 330 | 131 | 55 | 75 | 81 | 62 | 73 | 1097
  Male | 339 | 303 | 154 | 62 | 62 | 75 | 90 | 67 | 1152

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Serum Bactericidal Antibody Titers ≥1:5 After Receiving the Booster Dose of rMenB+OMV NZ Vaccination
Description: Immunogenicity was assessed in terms of the percentage of subjects as measured by serum bactericidal antibody titers ≥1:5 the lower limit of the two-sided 95% confidence interval (CI) was ≥75%, directed against N.meningitidis serogroup B reference strains H44/76-SL , NZ98/254, 5/99, one month after the booster (fourth) dose of meningococcal B vaccine with or without the concomitant Measles, Mumps, Rubella, Varicella (MMRV) vaccine in toddlers who were previously vaccinated with three doses of Meningococcal B vaccine.
Time Frame: one month after the booster (fourth) dose
Population: The analysis was done on Per Protocol (PP) population - subjects who received all doses of vaccine in parent & present study, provided evaluable serum samples at 1 month after booster dose or 1 month after 2nd dose, blood draw at 1 month after 3rd injection at 6 months in parent & visit 1 blood draw in present study, had no major protocol violation
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 12B12M (1a) | 12B13M (1b)
Number analyzed (Participants) | 211 | 215
Percentages of subjects
  Strain 44/76-SL (Baseline) (N=211, 215) | 81 [75 to 86] | 82 [77 to 87]
  One month after booster (N=210, 212) | 100 [98 to 100] | 100 [98 to 100]
  Strain 5/99 (Baseline) (N=210, 213) | 98 [95 to 99] | 100 [97 to 100]
  One month after booster (N=209, 212) | 100 [98 to 100] | 100 [98 to 100]
  Strain NZ98/254 (Baseline) (N=211, 215) | 19 [14 to 25] | 24 [19 to 30]
  One month after booster (N=211, 213) | 97 [93 to 99] | 94 [90 to 97]

2. Secondary Outcome: Percentages of Subjects With Antibody Response After Receiving the MMRV Vaccination
Description: Immunogenicity was assessed to demonstrate non-inferiority in terms of percentages of subjects as measured by antibody responses against MMRV vaccine when given concomitantly with the booster (fourth) dose of rMenB+OMV NZ vaccine at 12 months of age when compared to MMRV vaccine when given alone.
  The specified cut-off levels for the vaccine antigens : for measles antigen is ≥255mIU/mL, Mumps antigen is ≥10 Enzyme Linked Immunosorbent Assay(ELISA) Antibody(Ab) units, Rubella antigen is ≥10 IU/mL, Varicella antigen is ≥1.25 glycoprotein (gp) ELISA units/ml (seroconversion) and varicella antigen is ≥5 gp ELISA units/ml (seroprotection.
Time Frame: one month after booster (fourth) dose
Population: This analysis was done on Per Protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- 12B12M (1a): Previously in the parent study subjects had received three doses of rMenB+OMV NZ and routine vaccine at 2, 4 and 6 months of age, respectively. These subjects received a booster (fourth) dose at 12 months of age concomitantly with one dose of MMRV vaccine.
- 12M13B15B (2a): Previously in the parent study subjects had received only routine vaccine at 2, 4 and 6 months of age respectively. These subjects received MMRV vaccine at 12 months of age and two catch-up doses of rMenB+OMV NZ at 13 and 15 months of age in the present study.
Arm/Group | 12B12M (1a) | 12M13B15B (2a)
Number analyzed (Participants) | 163 | 156
Percentages of subjects
  Measles strain Schwarz≥255mIU/mLBaselineN=152,147 | 0 [0 to 2] | 0 [0 to 2]
  2 months after MMRV vaccine (N=151,146) | 98 [94 to 100] | 99 [96 to 100]
  Mumps(strain RIT4385)≥10 U/mL(Baseline)(N=157,152) | 0 [0 to 2] | 0 [0 to 2]
  2 months after MMRV vaccine (N=156, 151) | 96 [92 to 99] | 96 [92 to 99]
  Rubella (Wistar RA 27/3) ≥10 (Bas N=163,156) | 0 [0 to 2] | 0 [0 to 2]
  2 months after MMRV vaccine (N=162, 155) | 99 [96 to 100] | 100 [98 to 100]
  Varicella (Oka, ≥1.25), Bas (N=147,141) | 0 [0 to 2] | 0 [0 to 3]
  2 months after MMRV vaccine (N=146,140) | 97 [93 to 99] | 99 [95 to 100]
  Varicella (Oka, ≥5), Bas (N=147,141) | 0 [0 to 2] | 0 [0 to 3]
  VarII 2 months after MMRV vaccine (N=146, 140) | 79 [71 to 85] | 81 [73 to 87]
Statistical Analysis 1: Comparison: 12B12M (1a) vs 12M13B15B (2a); The immunogenicity in 12B12M (1a) group was considered non-inferior to that in group 12M13B15B (2a), if for the measles antigen (two months after the MMRV vaccine), the lower limit of the two-sided 95% CI for the difference in the percentages of subjects with antibody response greater than or equal to the specified cut-off level for Measles antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — The specified cut-off levels for the vaccine antigen measles is ≥255 mIU/mL to be greater than -10%; Percentage group difference = -1, 95% CI 2-sided [-5 to 2]
Statistical Analysis 2: Comparison: 12B12M (1a) vs 12M13B15B (2a); The immunogenicity in 12B12M(1a) group was considered non-inferior to that in group 12M13B15B(2a), if for the mumps antigen (two months after the MMRV vaccine), the lower limit of the two-sided 95% CI for the difference in the percentages of subjects with antibody response greater than or equal to the specified cut-off level for Mumps antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — The specified cut-off level for the vaccine antigen mumps is ≥10 Enzyme Linked Immunosorbent Assay(ELISA) Antibody (Ab) units to be greater than -10%; Percentage group difference = 0, 95% CI 2-sided [-5 to 5]
Statistical Analysis 3: Comparison: 12B12M (1a) vs 12M13B15B (2a); The immunogenicity in 12B12M(1a) group was considered non-inferior to that in group 12M13B15B (2a), if for the rubella antigen(two months after the MMRV vaccine), the lower limit of the two-sided 95% CI for the difference in the percentages of subjects with antibody response greater than or equal to the specified cut-off level for rubella antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — The specified cut-off level for the vaccine antigen rubella is ≥10 IU/mL to be greater than -10%; Percentage group difference = -1, 95% CI 2-sided [-4 to 1]
Statistical Analysis 4: Comparison: 12B12M (1a) vs 12M13B15B (2a); The immunogenicity in 12B12M(1a) group was considered non-inferior to that in group 12M13B15B (2a), if for the varicella antigen (two months after the MMRV vaccine), the lower limit of the two-sided 95% CI for the difference in the percentages of subjects with antibody response greater than or equal to the specified cut-off level for varicella antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — The specified cut-off value for the vaccine antigen varicella is ≥1.25 gpELISA units/mL to be greater than -10%; Percentage group difference = -1, 95% CI 2-sided [-6 to 3]
Statistical Analysis 5: Comparison: 12B12M (1a) vs 12M13B15B (2a); The immunogenicity in 12B12M (1a) group was considered non-inferior to that in group 12M13B15B (2), if for the varicella antigen (two months after the MMRV vaccine), the lower limit of the two-sided 95% CI for the difference in the percentages of the subjects with antibody response greater than or equal to the specified cut-off value for varicella antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — The specified cut-off level for the varicella vaccine antigen is ≥5 gp ELISA units/ml (seroprotection) to be greater than -10%; Percentage group difference = -2, 95% CI 2-sided [-11 to 7]

3. Secondary Outcome: The Geometric Mean Titers After Receiving the Booster Dose of rMenB+OMV NZ Vaccination
Description: The human serum bactericidal antibody (hSBA) titer responses, one month after receiving booster dose or rMenB+OMV NZ vaccination, are reported as geometric mean titers (GMTs).
Time Frame: one month after booster (fourth) vaccination.
Population: This analysis was done on PP population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 12B12M (1a) | 12B13M (1b)
Number analyzed (Participants) | 211 | 215
Titers
  Strain 44/76-SL (Baseline) | 11 [9.27 to 12] | 10 [9.11 to 12]
  1 Month after booster (N=210, 212) | 139 [123 to 156] | 119 [105 to 133]
  Strain 5/99 (N=210, 213) | 81 [71 to 93] | 81 [71 to 92]
  1 Month after booster (N=209, 212) | 1503 [1339 to 1686] | 1429 [1274 to 1603]
  Strain NZ98/254 (N=211, 215) | 2.07 [1.8 to 2.38] | 2.21 [1.92 to 2.55]
  1 Month after booster (N=211,213) | 39 [33 to 46] | 32 [27 to 37]

4. Secondary Outcome: Geometric Mean Titers at 12 Months of Age (Predose 4) After Previously Receiving the Three Doses of rMenB+OMV NZ (Persistence)
Description: The immunogenicity was assessed as the persistence of bactericidal antibodies at 12 months of age (pre-dose 4) who previously received three doses of rMenB+OMV NZ in the parent study as measured by hSBA GMTs directed against N meningitidis serogroup B reference strains H44/76, NZ98/254 and 5/99.
Time Frame: one month after third vaccination and pre dose fourth (booster) vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- 12B12M (1a): Previously in the parent study subjects had received three doses of rMenB+OMV NZ and routine vaccine at 2, 4 and 6 months of age, respectively. These subjets received a booster (fourth) dose at 12 months of age concomitantly with one dose of MMRV vaccine
- Men246: Combined groups of 1a and 1b who previously in the parent study subjects had received three doses of rMenB+OMV NZ and routine vaccine at 2, 4 and 6 months of age, respectively. These subjects received a booster (fourth) dose at 12 months of age and one dose of MMRV vaccine at 12 months (1a group) and at 13 months of age (1b) group in the present study.
- Routine246: Combined groups of 12M13B15B (2a) and 12M12B14B (2b) who previously received routine vaccine at 2, 4 an 6 months of age, respectively. These subjects received two catch-up doses of rMenB+OMV NZ at 13 and 15 months of age [12M13B15B (2a)]; 12 and 14 months [12M12B14B (2b)] in the parent study and one dose of MMRV vaccine at 12 months of age in both the groups in the present study.
Arm/Group | 12B12M (1a) | 12B13M (1b) | Men246 | Routine246
Number analyzed (Participants) | 139 | 133 | 272 | 51
Titers
  Strain 44/76-SL (Baseline) N=134, 131, 265,49 | 1.15 [1.05 to 1.27] | 1.15 [1.05 to 1.27] | 1.15 [1.08 to 1.24] | 1.14 [0.99 to 1.32]
  1 M after 3rd vac.in parent study N=139,133,272,51 | 91 [81 to 104] | 83 [73 to 94] | 87 [79 to 95] | 1.19 [1.07 to 1.33]
  Pre-Boodster vac.in present study N=139,133,272,51 | 11 [9 to 12] | 10 [8.7 to 12] | 10 [9.28 to 12] | 1.08 [0.99 to 1.17]
  Strain 5/99 (Baseline) N=132,129,261,49 | 1.13 [1.01 to 1.26] | 1.24 [1.11 to 1.39] | 1.18 [1.09 to 1.28] | 1.11 [1.01 to 1.22]
  1M after 3rd vac. in parent study N=139,133,272,51 | 615 [538 to 704] | 620 [540 to 712] | 617 [560 to 680] | 1 [1 to 1]
  Pre-Booster vac.in present study N=139,133,272,51 | 85 [72 to 100] | 79 [67 to 94] | 82 [73 to 92] | 1.03 [0.97 to 1.09]
  Strain NZ98/254 (Baseline) N=135,130,265,49 | 1.05 [0.98 to 1.13] | 1.12 [1.04 to 1.21] | 1.09 [1.03 to 1.15] | 1 [1 to 1]
  1M after 3rd vac. in parent study.N=139,132,271,52 | 12 [10 to 15] | 14 [12 to 17] | 13 [11 to 15] | 1.07 [0.94 to 1.21]
  Pre-booster vac in present study. N=139,132,271,52 | 2.04 [1.72 to 2.43] | 2.02 [1.69 to 2.42] | 2.03 [1.79 to 2.3] | 1 [1 to 1]

5. Secondary Outcome: Percentages of Subjects With Serum Bactericidal Antibody Titers ≥1:5 After Previously Receiving the Three Doses of rMenB+OMV NZ Vaccination (Persistence)
Description: Immunogenicity was assessed to evaluate the persistence in terms of percentages of subjects with hSBA titers ≥ 1:5, previously received three doses of rMenB+OMV NZ directed against N meningitidis serogroup B reference strains H44/76, NZ98/254 and 5/99.
Time Frame: One month post vaccination and pe-booster (fourth) dose vaccination
Population: The analysis was done on PP population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 12B12M (1a) | 12B13M (1b) | Men246 | Routine246
Number analyzed (Participants) | 139 | 133 | 272 | 51
Percentages of subjects
  44/76-SL Baseline in present studyN=134,131,265,49 | 3 [1 to 7] | 3 [1 to 8] | 3 [1 to 6] | 4 [0 to 14]
  1 M after 3rd vac in parent study.N=139,133,272,51 | 100 [97 to 100] | 99 [96 to 100] | 100 [98 to 100] | 0 [0 to 7]
  Pre-booster vac. in present study.N=139,133,272,51 | 81 [73 to 87] | 82 [74 to 88] | 81 [76 to 86] | 2 [0.05 to 10]
  5/99 Baseline in parent study N=132,129,261,49 | 4 [1 to 9] | 5 [2 to 10] | 4 [2 to 7] | 2 [0.052 to 11]
  1M after 3rd vac in parent study N=139,133,272,51 | 100 [97 to 100] | 99 [96 to 100] | 100 [98 to 100] | 0 [0 to 7]
  Pre-Boostervac.in present study N=139,133,272,51 | 98 [94 to 100] | 100 [97 to 100] | 99 [97 to 100] | 0 [0 to 7]
  NZ98/254 Baseline in parent study N=135,130,265,49 | 1 [0.019 to 4] | 4 [1 to 9] | 2 [1 to 5] | 0 [0 to 7]
  1 M after 3rd vac. in parent studyN=139,132,271,52 | 81 [74 to 87] | 85 [78 to 90] | 83 [78 to 87] | 2 [0.049 to 10]
  Pre-Booster vac in present study N=139,132,271,52 | 21 [14 to 29] | 20 [13 to 28] | 20 [16 to 26] | 0 [0 to 7]

6. Secondary Outcome: Geometric Mean Titers After Receiving the Booster Dose and Single Dose of rMen+OMV NZ Vaccination (Induction of Immunological Memory)
Description: The immunogenicity was assessed to demonstrate the induction of immunological memory in subjects who were previously received three doses of rMenB+OMV NZ as measured by SBA GMT response in comparison to the fourth dose of rMenB+OMV NZ at 12 months of age ( 12B12M(1a) group) to the response in subjects (12M12B14B 0 who received a single dose of rMenB+OMV NZ vaccine.
Time Frame: one month after booster (fourth) dose vaccination and pre-fourth dose vaccination
Population: This analysis was done on the PP population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- 12B12M (1a): Previously in the parent study subjects had received three doses of rMenB+OMV NZ and routine vaccine at 2, 4and 6 months of age, respectively. These subjects received a booster (fourth) dose at 12 months of age concomitantly with one dose of MMRV vaccine
- 12M12B14B (2b): Previously in the parent study subjects had received three doses of routine vaccine at 2, 4 and 6 months of age, respectively. These subjects received two catch-up doses of rMenB+OMV NZ at 12 and 14 months of age and one dose of MMRV vaccine was given concomitantly at 12 months of age in the present study
Arm/Group | 12B12M (1a) | 12M12B14B (2b)
Number analyzed (Participants) | 211 | 72
Titers
  44/76-SL (Baseline) (N=211, 71) | 11 [9.32 to 12] | 1.18 [0.96 to 1.46]
  1 M after Booster or 1st rMenB (N=210, 71) | 140 [123 to 159] | 15 [12 to 19]
  5/99 (Baseline) (N=210, 71) | 83 [73 to 93] | 1 [0.81 to 1.24]
  1 M after Booster or 1sr rMenB (N=209, 72) | 1538 [1337 to 1769] | 58 [46 to 74]
  NZ98/254 (Baseline) (N=211, 71) | 2.05 [1.83 to 2.31] | 1.03 [0.84 to 1.26]
  1M after Booster or 1st rMenB (N=211, 72) | 39 [34 to 46] | 4.18 [3.18 to 5.5]

7. Secondary Outcome: SBA GMTs After a Two-dose Catch-up Schedule or Two-dose Schedule
Description: The immunogenicity of a two-dose catch-up schedule of rMenB+OMV NZ given at 13 and 15 months (12M13B15B) or 12 and 14 months (12M12B14B) to naïve toddlers was assessed by SBA GMTs one month after the second dose.
Time Frame: One month after the second dose.
Population: The analysis was done on the SBA PP Catch-up population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- 12M12B14B (2b): Previously in the parent study subjects had received three doses of routine vaccine at 2, 4 and 6 months of age, respectively. These subjects received two catch-up doses of rMenB+OMV NZ at 12 and 14 months of age and one dose of MMRV vaccine given concomitantly at 12 months of age in the present study.
Arm/Group | 12M13B15B (2a) | 12M12B14B (2b)
Number analyzed (Participants) | 164 | 68
Titers
  Strain H44/76, Baseline (N=161,67) | 1.24 [1.15 to 1.35] | 1.22 [1.07 to 1.38]
  1 M after 2nd Vac. (N=163, 67) | 271 [237 to 310] | 248 [201 to 306]
  Strain 5/99, Baseline (N=160, 67) | 1.06 [1 to 1.13] | 1.03 [0.94 to 1.13]
  1 M after 2nd Vac. (N=164, 67) | 599 [520 to 690] | 627 [502 to 783]
  Strain NZ98/254, Baseline (N=162, 67) | 1.03 [0.98 to 1.07] | 1.03 [0.97 to 1.1]
  1M after 2nd Vac. (N=164, 68) | 43 [38 to 49] | 32 [26 to 40]

8. Secondary Outcome: Percentages of Subjects With SBA Titers ≥1:5 After a Two-dose Catch-up Schedule or Two-dose Schedule
Description: The immunogenicity of a two-dose catch-up schedule of rMenB+OMV NZ given at 13 and 15 months (12M13B15B) or 12 and 14 months (12M12B14B) to naïve toddlers was assessed as percentages of subjects with SBA titers ≥1:5 one month after the second dose.
Time Frame: One month after the second dose.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 12M13B15B (2a) | 12M12B14B (2b)
Number analyzed (Participants) | 164 | 68
Percentages of Subjects
  Strain H44/76, Baseline (N=161,67) | 5 [2 to 10] | 3 [0 to 10]
  1 M after 2nd Vac. (N=163, 67) | 100 [98 to 100] | 100 [95 to 100]
  Strain 5/99, Baseline (N=160, 67) | 1 [0 to 4] | 1 [0.038 to 8]
  1 M after 2nd Vac. (N=164, 67) | 100 [98 to 100] | 100 [95 to 100]
  Strain NZ98/254, Baseline (N=162, 67) | 1 [0.016 to 3] | 0 [0 to 5]
  1M after 2nd Vac. (N=164, 68) | 100 [98 to 100] | 96 [88 to 99]

9. Secondary Outcome: ELISA Geometric Mean Concentration Against Vaccine Antigen 287-953 One Month After the Fourth (Booster) Dose Given at 12 Months
Description: The immune response against vaccine antigen 287-953 was measured by ELISA, one month after the fourth (booster) dose given at 12 months of age (groups 12B12M (1a), 12B13M (1b).
Time Frame: One month after the fourth (booster) dose.
Population: The analysis was done on the SBA PP Booster population.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 12B12M (1a) | 12B13M (1b)
Number analyzed (Participants) | 213 | 216
IU/mL
  Baseline (N=212,216) | 390 [351 to 433] | 389 [349 to 434]
  1 M after Booster (N=213, 214) | 6225 [5571 to 6956] | 5608 [5111 to 6154]

10. Secondary Outcome: ELISA Geometric Mean Concentration Against Vaccine Antigen 287-953 After Two-dose Catch-up in Toddlers
Description: The immune response against vaccine antigen 287-953was measured by ELISA one month after the first dose and one month after the second dose of a two-dose catch-up regimens (12M13B15B and 12M12B14B) in toddlers.
Time Frame: One month after the first dose and one month after the second dose.
Population: The analysis was done on the SBA PP Catch-up population.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 12M13B15B (2a) | 12M12B14B (2b)
Number analyzed (Participants) | 165 | 68
IU/mL
  Baseline (N=162,66) | 20 [20 to 21] | 22 [19 to 24]
  1 M after 1st Vac. (N=162,64) | 113 [95 to 136] | 120 [88 to 164]
  1 M after 2nd Vac. | 5698 [5030 to 6454] | 7154 [5880 to 8704]

11. Secondary Outcome: Percentages of Subjects With Bactericidal Titers ≥ 1:5 (95% CI) Against Strain M10713 One Month After the Fourth (Booster) Dose Given at 12 Months
Description: The immune response was measured as percentages of subjects with SBA ≥ 1:5 (95% CI) against strain M10713, one month after the fourth (booster) dose given at 12 months of age (groups 12B12M (1a), 12B13M (1b).
Time Frame: One month after the fourth (booster) dose.
Population: The analysis was done on the SBA PP Booster population.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 12B12M (1a) | 12B13M (1b)
Number analyzed (Participants) | 19 | 27
Percentages of Subjects
  Pre-Booster Vac. | 84 [60 to 97] | 59 [39 to 78]
  1 Month After Booster | 100 [82 to 100] | 100 [87 to 100]

12. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Reactions During the 7 Days Following rMenB+OMV NZ Vaccination at 12 Months of Age
Description: Safety was assessed as the number of subjects who reported solicited local and systemic reactions from day 1 through day 7 after rMenB+OMV NZ vaccination administered at 12 months. For the safety analysis purpose, Groups 12B12M (1a) and 12B12M (3a) are combined as Group 12B12M and Groups 12B13M (1b) and 12B13M (3b) are combined as Group 12B13M.
Time Frame: From day 1 to day 7 after each rMenB+OMV NZ vaccination.
Population: Analysis performed on the Safety population.
Measure: Number; unit: Subjects
Groups:
- 12B12M: Combination of Groups 12B12M (1a) and 12B12M (3a).
- 12B13M: Combination of Groups 12B13M (1b) and 12B13M (3b).
Arm/Group | 12B12M_C (4a) | 12B13M_C (4b) | 12B12M | 12B13M
Number analyzed (Participants) | 152 | 138 | 765 | 789
Subjects
  Any local | 113 | 104 | 639 | 673
  MenB Tenderness | 97 | 80 | 546 | 563
  MenB Erythema | 78 | 81 | 504 | 539
  MenB Induration | 61 | 61 | 388 | 424
  MenB Swelling | 44 | 39 | 284 | 287
  Any systemic | 133 | 117 | 695 | 671
  Change Eat. Habits | 61 | 44 | 312 | 318
  Sleepiness | 64 | 60 | 362 | 355
  Vomiting | 9 | 10 | 54 | 36
  Diarrhea | 29 | 23 | 188 | 160
  Irritability | 89 | 75 | 560 | 540
  Unusual Crying | 48 | 48 | 327 | 294
  Rash | 8 | 7 | 57 | 56
  Rash Oth.to Fever | 6 | 0 | 31 | 0
  Rash Urt.to Fever | 2 | 0 | 18 | 0
  Rash Oth.to Doc. | 6 | 0 | 35 | 0
  Rash Urt.to Doc. | 2 | 0 | 23 | 0
  Gland Swelling | 4 | 0 | 12 | 0
  Gland Par.to Doc. | 0 | 0 | 0 | 0
  Gland Sal.to Doc. | 0 | 0 | 0 | 0
  Med. Att. Fever | 3 | 4 | 8 | 13
  Fever ( ≥ 38C ) | 87 | 74 | 356 | 325
  Antipyretic Med. Used | 79 | 69 | 436 | 406

13. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Reactions During the 7 Days Following Two-dose Catch-up Schedules of rMenB+OMV NZ Vaccination
Description: Safety was assessed as the number of subjects who reported solicited local and systemic reactions from day 1 through day 7 after rMenB+OMV NZ vaccination administered with a two-dose catch-up schedules (groups 12M13B15B and 12M12B14B).
Time Frame: From day 1 to day 7 after each rMenB+MV NZ vaccination.
Population: Analysis performed on the Safety population.
Measure: Number; unit: Subjects
Arm/Group | 12M13B15B (2a) | 12M12B14B (2b)
Number analyzed (Participants) | 284 | 117
Subjects
  Any local (1st vacc) | 211 | 92
  Any local (2nd vacc) | 212 | 90
  MenB Tenderness (1st vacc) | 158 | 67
  MenB Tenderness (2nd vacc) | 181 | 78
  MenB Erythema (1st vacc) | 173 | 79
  MenB Erythema (2nd vacc) | 159 | 70
  MenB Induration (1st vacc) | 111 | 57
  MenB Induration (2nd vacc) | 115 | 53
  MenB Swelling (1st vacc) | 81 | 36
  MenB Swelling (2nd vacc) | 83 | 33
  Any systemic (1st vacc) | 216 | 104
  Change Eat. Habits (1st vacc) | 96 | 44
  Any systemic (2nd vacc) | 224 | 99
  Change Eat. Habits (2nd vacc) | 83 | 43
  Sleepiness (1st vacc) | 110 | 55
  Sleepiness (2nd vacc) | 106 | 48
  Vomiting (1st vacc) | 14 | 2
  Vomiting (2nd vacc) | 8 | 3
  Diarrhea (1st vacc) | 41 | 34
  Diarrhea (2nd vacc) | 41 | 25
  Irritability (1st vacc) | 168 | 82
  Irritability (2nd vacc) | 153 | 73
  Unusual Crying (1st vacc) | 80 | 41
  Unusual Crying (2nd vacc) | 74 | 42
  Rash (1st vacc) | 13 | 9
  Rash (2nd vacc) | 10 | 4
  Rash Oth.to Fever (1st vacc) | 0 | 0
  Rash Oth.to Fever (2nd vacc) | 0 | 0
  Rash Urt.to Fever (1st vacc) | 0 | 0
  Rash Urt.to Fever (2nd vacc) | 0 | 0
  Rash Oth.to Doc. (1st vacc) | 0 | 0
  Rash Oth.to Doc. (2nd vacc) | 0 | 0
  Rash Urt.to Doc. (1st vacc) | 0 | 0
  Rash Urt.to Doc. (2nd vacc) | 0 | 0
  Gland Swelling (1st vacc) | 0 | 1
  Gland Swelling (2nd vacc) | 0 | 0
  Gland Par.to Doc. (1st vacc) | 0 | 0
  Gland Par.to Doc. (2nd vacc) | 0 | 0
  Gland Sal.to Doc. (1st vacc) | 0 | 0
  Gland Sal.to Doc. (2nd vacc) | 0 | 0
  Med. Att. Fever (1st vacc) | 0 | 1
  Med. Att. Fever (2nd vacc) | 2 | 2
  Fever (≥ 38C) (1st vacc) | 103 | 54
  Fever (≥ 38C) (2nd vacc) | 97 | 50
  Antipyr. Med. Used (1st vacc) | 119 | 67
  Antipyretic Med. Used (2nd vacc) | 107 | 58

14. Secondary Outcome: Number of Subjects Reporting Solicited Local Reactions During the 7 Days Following MMRV Vaccination at 12 Months of Age
Description: Safety was assessed as the number of subjects who reported solicited local reactions from day 1 through day 7 after the MMRV vaccination concomitantly with rMenB+OMV NZ at 12 months of age (groups 12B12M, 12M12B14B, 12B12M_C) or after MMRV vaccination alone without rMenB+OMV NZ at 12 months (Group 12M13B15B). For the safety analysis purpose, Groups 12B12M (1a) and 12B12M (3a) are combined as Group 12B12M.
Time Frame: From day 1 to day 7 after MMRV vaccination.
Population: Analysis performed on the Safety population.
Measure: Number; unit: Subjects
Arm/Group | 12M13B15B (2a) | 12M12B14B (2b) | 12B12M_C (4a) | 12B12M
Number analyzed (Participants) | 284 | 117 | 152 | 760
Subjects
  MMRV Tenderness | 56 | 39 | 68 | 353
  MMRV Erythema | 120 | 52 | 60 | 345
  MMRV Induration | 53 | 18 | 30 | 161
  MMRV Swelling | 31 | 11 | 28 | 122

15. Secondary Outcome: Number of Subjects Reporting Solicited Systemic Reactions During 8-28 Days Following MMRV Vaccination at 12 Months of Age
Description: Safety was assessed as the number of subjects who reported solicited systemic reactions from day 8 through day 28 after the MMRV vaccination concomitantly with rMenB+OMV NZ at 12 months of age (groups 12B12M, 12M12B14B, 12B12M_C) or after MMRV vaccination alone without rMenB+OMV NZ at 12 months (Group 12M13B15B). For the safety analysis purpose, Groups 12B12M (1a) and 12B12M (3a) are combined as Group 12B12M.
Time Frame: From day 8 to day 28 after MMRV vaccination.
Population: Analysis performed on the Safety population.
Measure: Number; unit: Subjects
Arm/Group | 12M13B15B (2a) | 12M12B14B (2b) | 12B12M_C (4a) | 12B12M
Number analyzed (Participants) | 284 | 117 | 152 | 760
Subjects
  Rash | 50 | 23 | 17 | 147
  Rash Oth.to Fever | 6 | 3 | 4 | 19
  Rash Urt.to Fever | 4 | 1 | 2 | 14
  Rash Oth.to Doc. | 3 | 1 | 3 | 10
  Rash Urt.to Doc. | 2 | 1 | 1 | 8
  Gland Swelling | 8 | 3 | 5 | 20
  Gland Par.to Doc. | 1 | 0 | 1 | 3
  Gland Sal.to Doc. | 1 | 0 | 1 | 5
  Med. Att. Fever | 19 | 6 | 15 | 54
  Fever ( ≥ 38C ) | 131 | 46 | 62 | 338
  Antipyretic Med. Used | 119 | 55 | 48 | 324

ADVERSE EVENTS:
Time Frame: All solicited and unsolicited Adverse Events (AEs) were collected from Day 1 to 7; serious AEs (SAEs), possibly or probably related, unrelated , medically attended and leading to premature withdrawal AEs were collected during the overall study period.
Groups:
- 12B12M: Previously in the parent study subjects had received three doses of rMenB+OMV NZ and routine vaccine at 2, 4 and 6 months of age,respectively. These subjects received a booster (fourth) dose at 12 months of age concomitantly with one dose of MMRV vaccine in the present study.
  This group is a combination of Groups 12B12M (1a) and 12B12M (3a) for safety data analysis purposes.
- 12B13M: Previously in the parent study subjects had received three doses of rMenB+OMV NZ and routine vaccine at 2, 4 and 6 months of age, respectively. These subjects received a booster (fourth) dose at 12 months and one dose of MMRV vaccine at 13 months of age in the present study.
  This group is a combination of Groups 12B13M (1b) and 12B13M (3b) for safety data analysis purposes.
Arm/Group | 12B12M | 12B13M | 12M13B15B (2a) | 12M12B14B (2b) | 12B12M_C (4a) | 12B13M_C (4b)
Serious Adverse Events (participants affected / at risk) | 28/765 | 40/789 | 27/284 | 9/117 | 7/152 | 2/139
Other Adverse Events (participants affected / at risk) | 754/765 | 760/789 | 282/284 | 116/117 | 145/152 | 132/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12B12M (N=765) | 12B13M (N=789) | 12M13B15B (2a) (N=284) | 12M12B14B (2b) (N=117) | 12B12M_C (4a) (N=152) | 12B13M_C (4b) (N=139)
Kawasaki's disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Strabismus correction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysplasia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vesicoureteric reflux (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Growth retardation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 6 (8) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exanthema subitum (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 4 (4) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12B12M (N=765) | 12B13M (N=789) | 12M13B15B (2a) (N=284) | 12M12B14B (2b) (N=117) | 12B12M_C (4a) (N=152) | 12B13M_C (4b) (N=139)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (45) | 46 (51) | 11 (13) | 7 (8) | 9 (15) | 11 (14)
Lymphadenopathy (Blood and lymphatic system disorders) | 29 (48) | 4 (4) | 13 (24) | 4 (6) | 8 (14) | 1 (1)
Somnolence (Nervous system disorders) | 362 (599) | 355 (569) | 178 (430) | 70 (154) | 64 (99) | 61 (91)
Crying (General disorders) | 327 (558) | 294 (467) | 132 (302) | 59 (140) | 48 (86) | 50 (83)
Injection site erythema (General disorders) | 549 (1891) | 539 (1326) | 213 (1018) | 94 (476) | 92 (316) | 82 (179)
Injection site induration (General disorders) | 419 (1392) | 424 (1188) | 165 (717) | 78 (325) | 67 (223) | 62 (159)
Injection site pain (General disorders) | 561 (1648) | 563 (1107) | 224 (759) | 89 (377) | 104 (329) | 81 (165)
Injection site swelling (General disorders) | 320 (874) | 287 (667) | 127 (418) | 53 (177) | 54 (166) | 40 (94)
Pyrexia (General disorders) | 511 (1136) | 356 (560) | 208 (584) | 85 (211) | 110 (256) | 80 (125)
Irritability (Psychiatric disorders) | 562 (1121) | 540 (996) | 226 (742) | 95 (300) | 89 (199) | 76 (142)
Eating disorder (Psychiatric disorders) | 313 (630) | 318 (582) | 156 (444) | 63 (152) | 61 (117) | 45 (84)
Diarrhoea (Gastrointestinal disorders) | 194 (342) | 171 (268) | 92 (215) | 48 (101) | 31 (57) | 25 (38)
Teething (Gastrointestinal disorders) | 13 (13) | 12 (13) | 20 (22) | 3 (3) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 56 (78) | 39 (53) | 38 (52) | 5 (7) | 11 (12) | 11 (21)
Rash (Skin and subcutaneous tissue disorders) | 178 (310) | 65 (104) | 78 (141) | 30 (61) | 22 (46) | 9 (13)
Bronchitis (Infections and infestations) | 60 (72) | 62 (78) | 38 (45) | 13 (16) | 12 (20) | 6 (9)
Conjunctivitis (Infections and infestations) | 46 (57) | 38 (42) | 22 (24) | 5 (5) | 7 (8) | 1 (2)
Ear infection (Infections and infestations) | 49 (60) | 59 (100) | 20 (37) | 14 (19) | 14 (18) | 6 (9)
Exanthema subitum (Infections and infestations) | 20 (21) | 27 (27) | 15 (15) | 3 (3) | 4 (4) | 2 (2)
Gastroenteritis (Infections and infestations) | 21 (22) | 25 (25) | 11 (11) | 2 (2) | 5 (6) | 7 (7)
Laryngitis (Infections and infestations) | 26 (26) | 27 (29) | 14 (19) | 7 (7) | 2 (2) | 6 (6)
Nasopharyngitis (Infections and infestations) | 49 (62) | 62 (81) | 37 (48) | 19 (28) | 3 (3) | 7 (7)
Otitis media (Infections and infestations) | 80 (121) | 79 (133) | 42 (56) | 10 (13) | 9 (10) | 7 (7)
Pharyngitis (Infections and infestations) | 38 (41) | 54 (64) | 19 (21) | 6 (6) | 7 (9) | 5 (6)
Rhinitis (Infections and infestations) | 30 (35) | 38 (43) | 26 (35) | 7 (7) | 3 (3) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 67 (83) | 59 (71) | 51 (66) | 11 (14) | 8 (12) | 9 (11)
Viral infection (Infections and infestations) | 33 (35) | 36 (38) | 23 (29) | 10 (11) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days